CLINICAL TRIAL: NCT05837312
Title: Pilot Test of Reconnecting to Internal Sensations and Experiences to Reduce Eating Pathology
Brief Title: Testing the Effects of RISE on Eating Pathology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, April Smith, Associate Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00001104
Record Dates: First submitted 2023-03-22; First posted 2023-05-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorder Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reconnecting to Internal Sensations and Experiences (Experimental): The interoceptive training consists of four 25-30 minute modules (plus 15-minutes worth of optional weekly practice) that focus on multiple aspects of interoception including: body awareness, body sensations and movement, eating, health and selfcare, emotional awareness, and understanding the self in relation to others. These modules are delivered weekly.
  Interventions: Behavioral: Reconnecting to Internal Sensations and Experiences

INTERVENTIONS:
Behavioral: Reconnecting to Internal Sensations and Experiences — Reconnecting to Internal Sensations and Experiences (RISE) is a novel, self-guided interoceptive intervention designed to be accessible and convenient. RISE is hosted on Qualtrics and accessed on any internet-enabled device. RISE consists of four interactive 30-minute modules: (1) Progressive Muscle Relaxation and Body Functionality, (2) Understanding, Noticing and Managing Emotions, (3) Self-care and Communication, and (4) Body Sensations. The training consists of a mix of audio clips, psychoeducation, self-guided reading, and interactive writing prompts. Intervention materials are separated by multiple free-response prompts so that participants can relate the materials to their own lives, practice the introduced skills, and problem-solve difficulties implementing the skills.

SUMMARY:
Interoception is the process of perceiving one's bodily sensations. Interoception is critical for survival and maintaining homeostasis, as it motivates sensation- and need-specific autonomic reflexes and adaptive behaviors (e.g., eating when hungry, terminating eating upon fullness, drinking when thirsty). Not all individuals have accurate interoceptive abilities. Individuals with eating disorders often have low perception of gastrointestinal, pain, and emotion sensations. Interoceptive dysfunction is believed to influence the development and maintenance of many forms of psychopathology. Identifying effective ways to restore accurate interoceptive processing is an important aim for clinical researchers. The goal of the present study is to continue to test the effectiveness of a training for interoceptive dysfunction that aims to reconnect individuals with eating disorders with their internal sensations, which is called, Reconnecting to Internal Sensations.

DETAILED DESCRIPTION:
There are individual differences in how well people are able to recognize interoceptive sensations. Research supports a role for impaired interoception in the etiology of eating disorders (EDs), with the idea being that individuals who are out of touch with hunger and/or satiety are more vulnerable to restrictive and binge eating behaviors, respectively. Researchers have connected interoceptive impairment to self-injurious behaviors more broadly, including both direct (i.e., non-suicidal self-injury and suicide attempts) and indirect (i.e., ED behaviors) forms. The investigators have found support for the supposition that impaired interoception-or bodily disconnect-allows people to inflict pain (whether that be through ED behaviors or self-injury) upon themselves, as it is much easier to harm something one is unattached to versus something one cares for. Thus, improving interoception (e.g., helping people connect better with their bodies) may improve ED outcomes. This project seeks to test an accessible, online intervention designed to improve interoception and thereby reduce ED symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an eating disorder
* Be a patient at the Louisville Center for Eating Disorders
* Above age 10

Exclusion Criteria:

*Under age 10

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness, Version 2 | Within one week of completing the intervention
  The Multidimensional Assessment of Interoceptive Awareness, Version 2 is 37-item scale that has 8 subscales that measure the ability to recognize and accurately identify emotions and physiological sensations. Each item is rated on a 0-5 Likert scale, thus total scores can range from 0-185. Higher scores indicate better interoceptive awareness.
Eating Disorder Inventory - Interoceptive Deficits Subscale | Within one week of completing the intervention
  10 item subscale assessing interoceptive deficits, including gastrointestinal interoception

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire | Within one week of completing the intervention
  The Eating Disorder Examination Questionnaire is a self-report assessment of eating disorder symptoms that assesses eating disorder behaviors (e.g., excessive exercise, binging, purging, fasting) and includes 4 subscales: weight concerns, shape concerns, restraint, and eating concerns. Items are rated on a 0 (No days) to 6 (Every day) scale. The global score is computed by summing the items and taking the mean, thus scores can range from 0-6. Higher scores indicate more eating pathology.

OTHER OUTCOMES:
Treatment Acceptability Questionnaire | Within one week of completing the intervention
  The Treatment Acceptability Questionnaire (TAQ) is a 6-item self-report assessment of the acceptability of the treatment. However in the current study the item pertaining to "How knowledgeable the psychologist is" will be removed as the intervention is delivered online; thus, the TAQ will be assessed with 5 items. Items are rated on a 1-7 Likert scale, and scores can range from 1-35. Higher scores indicate more treatment acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Louisville Center For Eating Disorders, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith AR, Forrest LN, Perkins NM, Kinkel-Ram S, Bernstein MJ, Witte TK. Reconnecting to Internal Sensation and Experiences: A Pilot Feasibility Study of an Online Intervention to Improve Interoception and Reduce Suicidal Ideation. Behav Ther. 2021 Sep;52(5):1145-1157. doi: 10.1016/j.beth.2021.02.001. Epub 2021 Feb 20. PMID 34452669
- [Background] Smith AR, Kinkel-Ram S, Grunwald W, George TS, Raval V. A Pilot Feasibility Study of Reconnecting to Internal Sensations and Experiences (RISE), a Mindfulness-Informed Intervention to Reduce Interoceptive Dysfunction and Suicidal Ideation, among University Students in India. Brain Sci. 2022 Feb 9;12(2):237. doi: 10.3390/brainsci12020237. PMID 35204000
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Mond JM, Hay PJ, Rodgers B, Owen C. Eating Disorder Examination Questionnaire (EDE-Q): norms for young adult women. Behav Res Ther. 2006 Jan;44(1):53-62. doi: 10.1016/j.brat.2004.12.003. PMID 16301014